CLINICAL TRIAL: NCT00643877
Title: A Prospective,Multi-Center,Randomized Control Trial of Preoperative Hepatic and Regional Arterial Chemotherapy(PHRAC) Using Oxaliplatin, Fluorodeoxyuridine(FUDR) and Mitomycin C(MMC) to Prevent Postoperative Liver Metastasis of Colorectal Cancer
Brief Title: Trial of Preoperative Hepatic and Regional Arterial Chemotherapy (PHRAC) to Prevent Postoperative Liver Metastasis of Colorectal Cancer
Acronym: PHRAC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Ruijin Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); First Affiliated Hospital of Zhejiang University (Other); Jiangyin People's Hospital (Other); Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Xujianmin, Zhongshan hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008-46
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasms; Regional; Liver; Neoplasm Metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Floxuridine; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Experimental): PHRAC was performed 7 days before surgery. Adjuvant chemotherapy using FOLFOX7 was done for 8 cycle with 28 days after surgery.
  Interventions: Procedure: Preoperative hepatic and regional arterial chemotherapy using oxaliplatin, MMC and FUDR
- A (No Intervention): Adjuvant chemotherapy using FOLFOX7 was done for 8 cycle with 28 days after surgery.
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: Preoperative hepatic and regional arterial chemotherapy using oxaliplatin, MMC and FUDR — PHRAC which included of two parts(common hepatic artery chemotherapy and main tumor supplying artery chemotherapy) was performed 7 days before surgery： common hepatic artery chemotherapy: FUDR 500mg, Oxaliplatin 50mg and MMC 10mg main tumor supplying artery chemotherapy: FUDR 500mg, Oxaliplatin 50mg and MMC 10mg
  Arms: B
Procedure: surgery — radical surgery only
  Arms: A

SUMMARY:
The purpose of this study is to investigate whether preoperative hepatic and regional arterial chemotherapy are able to prevent liver metastasis and improve overall survival in patients receiving curative colorectal cancer resection.

DETAILED DESCRIPTION:
We administered FUDR, MMC and Oxaliplatin as preoperative hepatic and regional arterial chemotherapy (PHRAC) to patients with Stage II or Stage III colorectal cancer without apparent liver metastasis based on a thorough preoperative evaluation. The study endpoints were disease-free survival, overall survival, and liver metastasis-free survival as evaluated by intent-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* age < 75 years with histologically proven adenocarcinoma of the colon or rectum
* no severe major organ dysfunction
* WHO performance status of 0 or 1
* no prior cancer therapy
* Stage II (T3-4, N0, M0) or Stage III (T0-4, N1-2, M0) disease (according to the 1997 revision of the International Union Against Cancer TNM staging system) as determined by a preoperative evaluation that included colonoscopy and an abdominal computed tomography (CT) scan

Exclusion Criteria:

* age >= 75
* severe major organ dysfunction
* WHO performance status of >1
* prior cancer therapy
* Stage I or Stage IV

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
5 years disease-free survival | 5 years after operation

SECONDARY OUTCOMES:
5 years overall survival and liver metastasis-free survival | 5 years after operation

CONTACTS AND LOCATIONS:
Overall Officials: jianmin xu, MD, Study Chair — department of general surgery, zhongshan hospital, fudan university
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

REFERENCES:
- [Derived] Zhu D, Xia J, Gu Y, Lin J, Ding K, Zhou B, Liang F, Liu T, Qin C, Wei Y, Ren L, Zhong Y, Wang J, Yan Z, Cheng J, Chen J, Chang W, Zhan S, Ding Y, Huo H, Liu F, Sun J, Qin X, Xu J. Preoperative Hepatic and Regional Arterial Chemotherapy in Patients Who Underwent Curative Colorectal Cancer Resection: A Prospective, Multi-center, Randomized Controlled Trial. Ann Surg. 2021 Jun 1;273(6):1066-1075. doi: 10.1097/SLA.0000000000004558. PMID 33214446